CLINICAL TRIAL: NCT06942390
Title: Topical Metfotmin Versus Topical Ketotifen (Alone or in Combination With Microneddling)in Melasma Treatment :Comparative Split Face Study
Brief Title: Topical Metformin Versus Topical Ketotifen in Melasma Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Khaled AbdElAziz, resident at the dermatology department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Melasma treatment
Record Dates: First submitted 2025-03-26; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Metformin; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Micro-Needling Combined with Topical Treatments (Experimental): This arm involves 51 patients receiving four sessions of micro-needling across their entire face at four-week intervals. After micro-needling, topical ketotifen is applied to one half of the face and topical metformin to the other half. Between sessions, patients continue daily application of both treatments.
  Interventions: Device: Micro-Needling Combined with ketofin and metformin
- topical Treatments Alone (Experimental): This arm includes 51 patients receiving daily applications of topical ketotifen on one half of their face and topical metformin on the other half without undergoing micro-needling sessions.
  Interventions: Drug: ketofin and metformin Alone

INTERVENTIONS:
Device: Micro-Needling Combined with ketofin and metformin — After micro-needling, topical ketotifen is applied to one half of the face and topical metformin to the other half. Between sessions, patients continue daily application of both treatments.
  Arms: Micro-Needling Combined with Topical Treatments
Drug: ketofin and metformin Alone — This arm includes 51 patients receiving daily applications of topical ketotifen on one half of their face and topical metformin on the other half without undergoing micro-needling sessions.
  Other Names: topical treatments
  Arms: topical Treatments Alone

SUMMARY:
The study aims to evaluate and compare the efficacy and safety of a new formulation of topical metformin (nanoparticles) versus topical ketotifen (nanoparticles), both alone and combined with micro-needling, for the treatment of melasma. It is a double-blinded, randomized, split-face controlled clinical study involving 102 female patients diagnosed with bilateral melasma.

DETAILED DESCRIPTION:
This research investigates the therapeutic effects of two nanoparticle-based topical treatments-metformin and ketotifen-on melasma. The study employs a split-face design where each patient receives different treatments on each half of their face. Patients are divided into two groups:

Group 1: Undergoes micro-needling sessions for the entire face, followed by the application of topical ketotifen on one half and topical metformin on the other half.

Group 2: Receives only topical applications of ketotifen on one half of the face and metformin on the other half without micro-needling.

The study includes detailed pre-procedure preparation (cleaning and anesthetizing the face) and post-procedure care (application of SPF 50+ sunblock). Clinical assessments include photographic documentation, H-MASI and mH-MASI scoring for melasma severity, patient satisfaction surveys, MELASQOL questionnaires to assess quality-of-life impacts, and monitoring for side effects. Assessments are conducted at baseline, monthly during treatment, and one month after the final session.

ELIGIBILITY:
Inclusion Criteria:

* Female adults of 18 years and above with bilateral melasma .
* Clinical diagnosis of melasma.
* Mental capacity to give informed consent.

Exclusion Criteria:

* Pregnant or nursing women.
* Current use of hormonal birth control medication or any hormonal therapy.
* Current or previous treatment by depigmenting agents within 3 months
* History of laser or MN to the face within 3 months of study enrollment.
* Patients with poor wound healing, recurrent herpes simplex and current skin infection (facial warts, molluscum contagiosum) and history of hypertropic scar/keloids.
* Photosensitivity.
* Patients with unrealistic expectations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Melasma Severity Index (MASI) Score | 1 month
  Measurement of changes in MASI score from baseline to the end of treatment (1 month). MASI is a validated tool used to assess the severity and area of melasma pigmentation, with lower scores indicating improvement.The Melasma Area and Severity Index (MASI) quantifies melasma severity using a 0-48 scale, where 0 = no melasma and 48 = maximum severity

CONTACTS AND LOCATIONS:
Overall Officials: Radwa Bakr, Assistant professor, Study Director — Assiot university

IPD SHARING:
Plan to Share IPD: No